CLINICAL TRIAL: NCT05746845
Title: RESEPTOR 5-HT7 : Interest of the 5-HT7 Serotonin Receptor as a Biomarker in Multiple Sclerosis
Brief Title: Implication of 5-HT7 Receptor in Inflammatory Mechanisms in Multiple Sclerosis
Acronym: RESEPTOR 5-HT7
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2021-07
Record Dates: First submitted 2023-01-25; First posted 2023-02-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Multiple Sclerosis
Keywords: Multiple sclerosis; Serotonin; 5-HT7 receptor; Inflammation; Lymphocytes; Monocytes; Cytokines
MeSH Terms: conditions — Multiple Sclerosis; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy individuals: Group 1: Healthy individuals, so-called "control" donors whose blood samples will be collected from the EFS (French Blood Establishment)
  Interventions: Biological: Blood sample
- Stable MS patients treated with high efficacy treatment: Group 2: Stable MS patients without inflammatory activity of the disease treated with high efficacy treatment (Natalizumab or Ocrelizumab)
  Interventions: Biological: Blood sample
- Stable MS patients treated with moderately effective treatment: Group 3: Stable MS patients without inflammatory disease activity treated with moderately effective treatment (Teriflunomide or Fumarate)
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood sampling will be done on three groups:
  Group 1: Healthy volunteers, so-called "control" donors whose blood samples will be ordered from the EFS (French Blood Establishment) Group 2: Stable MS patients without inflammatory activity of the disease treated with high efficacy treatment (Natalizumab or Ocrelizumab) Group 3: Stable MS patients without inflammatory disease activity treated with moderately effective treatment (Teriflunomide or Fumarate)

SUMMARY:
Multiple Sclerosis is a chronic autoimmune disease associated with inflammatory response harmful for the Central Nervous System. Immunological imbalance is involved with Th1 and Th17 cells in correlation with a disturbance of regulators mechanisms as Treg cells. Despite years of research, the mechanisms involved remain unclear.

Serotonin (5-HT) seems to be play an essential role in developing CNS inflammatory diseases and in particular in MS. Indeed, several studies have shown the anti-inflammatory potential of this neurotransmitter and also its vulnerability in inflammatory context. Moreover, a recent study has shown that 5-HT can reduced CD4 T cells proliferation and pro-inflammatory cytokines released in vitro. Interestingly, treatment, treatment with SSRIs (selective serotonin reuptake inhibitor) in an animal model of MS, on Experimental Autoimmune Encephalomyelitis, was shown to improve the clinical score and promote remission of the disease.

Among serotonin receptors, the 5-HT7 receptor, can be considered as an interesting target to treat neurological disorders associated with inflammatory context. Present in humans and mice, this receptor is expressed on the surface of a large number of cells, such as T-lymphocytes, macrophages, dendritic cells as well as on cells of CNS such as neurons, astrocytes and microglia.

Given the importance of the positive cells for 5-HT7 receptor, in the inflammatory context observed in multiple sclerosis, the investigators propose to study the receptor expression in blood samples from multiple sclerosis patient.

DETAILED DESCRIPTION:
In a previous translational study (5-HT SEP), the expression modulation of 5-HT7 receptor in function of immunological context was investigated, in different group of MS patients:

* Group 1: MS patients with an acute relapse
* Group 2: MS stable patients treated with Natalizumab
* Group 3: Healthy people (from Etablissement Français du Sang) From blood cells of different groups of individuals, the investigators determined the percentage and intensity of expression of the receptor on circulating lymphocytes by flow cytometry.

The investigators demonstrated in this first study that the 5-HT7 receptor is mainly expressed on the surface of B lymphocytes compared to T lymphocytes.

Interestingly, while the percentage of T lymphocytes (CD4+, CD8+) remained unchanged between the 3 groups, the investigators observed that the expression of R5-HT7 on the surface of the T lymphocyte subpopulations (Th1, Th2, Th17 and Treg), is significantly increased in the blood of MS patients treated with Natalizumab compared to healthy individuals and MS patients in relapse.

Considering litterature data and our preliminary results showing the therapeutic potential of 5-HT7R ligand in animal models of MS as well as the upregulation of 5-HT7 expression in NTZ-treated patients (5-HTSEP study), the investigators wish to go further with these investigations. The main objective of this new translational study is to demonstrate the interest of the 5-HT7 serotonin receptor as a biomarker in the therapeutic monitoring of patients suffering from Multiple Sclerosis.

The investigators first want to know if the increase in the expression of R5-HT7 on the surface of lymphocyte populations in stable MS patients is due specifically to Natalizumab treatment or if other treatments would also induce a similar effect. To answer this question, the investigators will study the expression of the receptor not only on the surface of lymphocyte cells but also on the surface of monocytes, NK cells and polymorphonuclear cells (cells not investigated in the first 5-HTSEP study) in three groups of individuals:

* Group 1: Healthy individuals, so-called "control" donors whose blood samples will be collected from the EFS (French Blood Establishment)
* Group 2: Stable MS patients without inflammatory activity of the disease treated with high efficacy treatment (Natalizumab or Ocrelizumab)
* Group 3: Stable MS patients without inflammatory disease activity treated with moderately effective treatment (Teriflunomide or Fumarate)

Group 1 (healthy volunteers) is a control group necessary for the smooth running of the study and the interpretation of the results.

For group 2, the Natalizumab treatment has already been investigated during the previous 5-HTSEP study. This new study will make it possible to 1) compare the expression/activity of the receptor in the three groups 2) check the reproducibility of the results compared to the previous study 3) evaluate any variations linked to the temporality of the treatment with 2 blood samples, a first before injection of Natalizumab, a second 14 days later. Indeed, unlike the 5-HTSEP study, where a single sample 1 month after injection of Natalizumab was analysed, the investigators wish to take these two samples, in order to carry out a longitudinal study making it possible to observe the evolution of the expression of the 5-HT7 receptor as a function of the temporality of the treatment.

Group 3 will assess whether other treatments (teriflunomide or fumarate) can induce an effect similar to that observed after Natalizumab treatment which is associated with an increase of R5-HT7 expression on the surface of lymphocyte populations in stable MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged between 18 and 50 years old,
* With multiple sclerosis already diagnosed and fulfilling the modified Mc Donald criteria
* Stable (no relapse in the last 6 months and MRI less than a year old, with no new lesions) and with at least 1 year of treatment with Natalizumab, Ocrelizumab, Teriflunomide or Fumarate
* Subject medically fit to give a maximum of 50 ml of extra whole blood
* Patient having given their consent to participate in the study

Exclusion Criteria:

* HIV serology known or discovered during the present episode
* Demented patient
* Patient treated with corticosteroids in the last month
* Non-affiliated person or non-beneficiary of a social security scheme
* Uncooperative patient
* Patient under legal protection, guardianship or curatorship
* Pregnant or breastfeeding women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Group 1: Healthy individuals, so-called "control" donors whose blood samples will be collected from the EFS (French Blood Establishment) Group 2: Stable MS patients without inflammatory activity of the disease under high efficacy treatment (Natalizumab or Ocrelizumab) Group 3: Stable MS patients without inflammatory disease activity under moderately effective treatment (Teriflunomide or Fumarate)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
5-HT7 receptor expression on circulating cells | Day 1
  using the flow cytometry technique, on whole blood, we will perform immunophenotyping in order to determine the fluorescence intensity of cells positive for the receptor (5-HT7+ cells) (B, T and NK lymphocytes, monocytes, and polynuclear cells) in the different groups of individuals.

SECONDARY OUTCOMES:
Expression of the 5-HT7 receptor after positive selection of different cell populations from PBMC | Day 15
  After Ficoll gradient, a part of PBMC (peripheral blood mononuclear cells) will be used to study the expression of the 5-HT7 receptor by positive selection of different cell populations (B lymphocytes, T lymphocytes, monocytes) using magnetic beads. Measurements of mRNA expression (R5-HT7, 5-HT synthesis enzyme, 5-HT transporter as well as markers of inflammation/autophagy) will be carried out by RT-qPCR.
Expression of the different isoforms of the 5-HT7 receptor on PBMC | Day 15
  In humans, there are three isoforms, obtained by alternative splicing, of the receptor, 5-HT7a, 5-HT7b, 5-HT7d, which differ according to the length of their C-terminal part. To date, no differences between these isoforms from a pharmacological and transductional point have been described. However, it would be interesting to quantify them by RTqPCR using mRNA from total PBMCs and then mRNA from the main populations of PBMCs, obtained by magnetic sorting, in order to assess their proportion.
Functional activity of the 5-HT7 receptor on PBMC: protein studies | Day 15
  A part of PBMCs (peripheral blood mononuclear cells) will be cultured and stimulated under different conditions: LPS stimulation (lipopolysaccharide), PHA stimulation (phytohemagglutinin), both stimulation LPS+PHA or with agonists and antagonists, as well as biased ligands of the receptor. After stimulation, cell supernatants will be collected in order to performed protein assays by ELISA technique (Enzyme-Linked Immunosorbent Assay). We want to measure the production of pro and anti-inflammatory cytokines (IL-1β, IL-4, TNFα, IL6, IL-17, IFN-γ and IL-10 and others based on literature data) to evaluate the effect of the different conditions of stimulation of PBMCs from the 3 group of patients
Functional activity of the 5-HT7 receptor on PBMC: mRNA expression studies | Day 15
  A part of PBMCs (peripheral blood mononuclear cells) will be cultured and stimulated under different conditions: LPS stimulation (lipopolysaccharide), PHA stimulation (phytohemagglutinin), both stimulation LPS+PHA or with agonists and antagonists, as well as biased ligands of the receptor. After stimulation, mRNA expression measurements (R5-HT7, 5-HT synthesis enzyme, 5-HT transporter as well as markers of inflammation/autophagy) will be performed by qPCR.
Relationship between Multiple sclerosis treatment on inflammation and serotonin production in serum | Day 15
  After Ficoll gradient, serum will be collected. Serotonin levels will be measured and different pro and anti-inflammatory mediators like IL-1β, IL-4, TNFα, IL6, IL8, IL-17, IFN-γ, GM-CSF and IL-10 and others based on literature data, will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Maud PALLIX-GUYOT, Dr, Principal Investigator — CHU Orleans
Locations (1):
- CHU Orléans, Orléans, France

REFERENCES:
- [Result] Sacramento PM, Monteiro C, Dias ASO, Kasahara TM, Ferreira TB, Hygino J, Wing AC, Andrade RM, Rueda F, Sales MC, Vasconcelos CC, Bento CAM. Serotonin decreases the production of Th1/Th17 cytokines and elevates the frequency of regulatory CD4+ T-cell subsets in multiple sclerosis patients. Eur J Immunol. 2018 Aug;48(8):1376-1388. doi: 10.1002/eji.201847525. Epub 2018 Jun 6. PMID 29719048
- [Result] Yuan XQ, Qiu G, Liu XJ, Liu S, Wu Y, Wang X, Lu T. Fluoxetine promotes remission in acute experimental autoimmune encephalomyelitis in rats. Neuroimmunomodulation. 2012;19(4):201-8. doi: 10.1159/000334095. Epub 2012 Mar 21. PMID 22441536